CLINICAL TRIAL: NCT03026686
Title: Postpartum Preeclampsia Readmission
Brief Title: Postpartum Readmission
Status: Terminated | Type: Observational
Why Stopped: Insufficient personel
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, Principal investigator, St. Louis University
Other Study IDs: 24998
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Postpartum Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- readmit: women who were re-admitted in the post partum period for a hypertensive disorder
- Controls: women with similar risk factors but did not require readmission

SUMMARY:
This is a retrospective chart review of women who labored and delivered in a single health care center. From that large group the investigators will evaluate women who were re-admitted in the post partum period for a hypertensive disorder. The study will also look at "Controls," a group of women with similar risk factors but did not require readmission.

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-specific multisystem disorder of unknown etiology. The disorder affects approximately 10 percent of pregnancies worldwide constituting one of the greatest causes of maternal and perinatal morbidity and mortality worldwide. (1) Preeclampsia is defined by the new onset of elevated blood pressure after 20 weeks of gestation. It is considered severe if blood pressure is increased substantially or symptoms of end-organ damage (including fetal growth restriction) occur. There is no single reliable, cost-effective screening test for preeclampsia, and there are no well-established measures for primary prevention. Management before the onset of labor includes close monitoring of maternal and fetal status. Management during delivery includes seizure prophylaxis with magnesium sulfate and, if necessary, medical management of hypertension. Delivery remains the ultimate treatment.

Preeclampsia leads to eclampsia. Symptoms of preeclampsia include: weight gain, headaches, right upper quadrant pain, swelling of hands and feet, and vision problems Symptoms of eclampsia include: muscle aches and pains, seizures, severe agitation, unconsciousness

Current obstetric treatment in the United States has resulted in a shift of eclampsia toward the postpartum period, with most cases being seen as late post partum. During the post partum period a patient's blood pressure peaks around 3-6 days post delivery, however most patients are discharged home by 48 hours. This results in re-admission to the hospital for some women. The investigator's goal is to review and evaluate women who have been readmitted for a preeclampsia or eclampsia episode during the post partum period to assess if there are preceding signs or symptoms leading to her re admission.

ELIGIBILITY:
Inclusion Criteria:

* Women who labored and delivered at a single hospital Readmitted (within 6 weeks post partum (PP) or less)to the hospital for hypertension disorder, with or without hypertension (HTN in pregnancy), gestational hypertension (gHTN), pre eclampsia (PreE), severe pre eclampsia (sPreE), HELLP ("HELLP" is an abbreviation of the three main features of the syndrome: Hemolysis. Elevated Liver enzymes. Low Platelet count.).

Controls Group with PreE, not readmitted or No PreE

Exclusion Criteria:

* Hospital readmission for other complications.

Ages: 14 Years to 55 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Women postpartum who are re-admitted for hypertension disorders
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
hypertension | 1 year
  compare these two groups during the antepartum period, labor, delivery and post partum course for possible preceding signs (blood pressures) of those at risk for re admission for hypertensive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No